CLINICAL TRIAL: NCT06800638
Title: Clinical Presentation, Diagnostic Approaches, Pathophysiology, and Management of Retinal Pseudo-Holes: a Comprehensive Synthesis of 35 Peer-Reviewed Studies
Brief Title: Comprehensive Review of Retinal Pseudo-Holes: Clinical Presentation, Diagnosis, Pathophysiology, and Management
Status: Completed | Type: Observational
Sponsor: Mohammad Reza Tokhmehchi (Other)
Responsible Party: Sponsor-Investigator, Mohammad Reza Tokhmehchi, Director, Hamadan University of Medical Science
Organization: Hamadan University of Medical Science (Other)
Other Study IDs: IR.GUMS.REC.1400.134
Record Dates: First submitted 2025-01-12; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Epiretinal Membrane; Age-related Disease; Idiopathic ERM
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retinal pseudo-holes (RPH) are macular abnormalities that mimic macular holes (MH) but lack full-thickness retinal disruption. This systematic review, based on 35 studies, explores their clinical presentation, diagnosis, pathophysiology, and management.

Diagnosis: Differentiating RPH from MH is challenging due to overlapping symptoms such as central scotomas and visual distortion. Optical coherence tomography (OCT) has become the gold standard for diagnosis, surpassing older imaging techniques like fundus photography and fluorescein angiography. OCT provides detailed, non-invasive imaging that helps identify RPH's hallmark feature: a foveal depression without retinal break.

Pathophysiology: RPH is primarily caused by mechanical forces exerted on the macula by epiretinal membranes (ERM) and vitreomacular traction (VMT). These forces distort the retina, creating a pseudo-hole. Risk factors include aging, high myopia, trauma, and diabetes.

Management: Many RPH cases are managed conservatively with regular monitoring, as the condition often remains stable. Surgical intervention, such as pars plana vitrectomy (PPV) with membrane peeling, is reserved for symptomatic cases with significant visual impairment. Surgery has shown promising outcomes, with most patients experiencing improved visual acuity.

Research Needs: Further studies are needed to explore the long-term outcomes of RPH, identify factors predicting progression to MH, and assess the utility of advanced imaging techniques like OCT angiography in improving diagnosis and monitoring.

This review underscores the importance of accurate differentiation between RPH and MH to ensure appropriate management and avoid unnecessary treatments.

DETAILED DESCRIPTION:
This is a REVIEW study on Retinal pseudo-holes.

ELIGIBILITY:
Inclusion Criteria:

* Studies that directly addressed retinal pseudo-holes, their clinical presentation, diagnostic modalities, pathophysiology, or treatment.
* Peer-reviewed clinical trials, case reports, observational studies, and reviews.
* Studies that utilized OCT or other imaging techniques (such as fluorescein angiography or fundus photography) to diagnose retinal pseudo-holes.
* Studies that were published in English and provided full-text access.

Exclusion Criteria:

* Studies that did not specifically focus on retinal pseudo-holes but instead dealt with other retinal conditions (e.g., full-thickness macular holes, retinal detachment).
* Studies that were not peer-reviewed (e.g., conference abstracts, opinion pieces).
* Non-English language studies or those without available full texts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 35
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | up to 12 weeks
  Measuring retinal thickness using Optical Coherence Tomography (OCT) to assess structural changes associated with the severity of the epiretinal membrane. Unit of Measure: Micrometers (µm)

SECONDARY OUTCOMES:
Visual Acuity | up to 10weeks
  Evaluating patients' visual acuity using the LogMAR scale to determine the functional impact of the epiretinal membrane on vision. Unit of Measure: LogMAR (logarithm of the minimum angle of resolution)

CONTACTS AND LOCATIONS:
Locations (1):
- Hamadan University of Medical Sciences, Hamadan, Iran